CLINICAL TRIAL: NCT05268796
Title: Randomized Controlled Trial of Telehealth-Enabled Versus In-Person Parent-Mediated Behavioral Treatment for Challenging Behaviors in Children With Autism Spectrum Disorder
Brief Title: Telehealth-Enabled Versus In-Person Parent-Mediated Behavioral Treatment for Challenging Behaviors in Children With ASD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Behavior Change Institute (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott Hall, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR210221
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person treatment (Active Comparator)
  Interventions: Behavioral: Behavior therapy
- Telehealth-enabled treatment (Active Comparator)
  Interventions: Behavioral: Behavior therapy
- Psychoeducation (Placebo Comparator)
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Behavior therapy — Caregivers will be coached either in-person or via telehealth to implement function-based behavioral treatment in 1-hour sessions each week with their child over 12 weeks.
  Arms: In-person treatment; Telehealth-enabled treatment
Other: Psychoeducation — Caregivers will complete online education modules in 1-hour sessions each week over 12 weeks.
  Arms: Psychoeducation

SUMMARY:
The purpose of the research is to determine whether parent-mediated behavior therapy for challenging behavior commonly displayed by children with autism spectrum disorder (ASD) can be as effective when delivered via telehealth as when delivered in-person.

ELIGIBILITY:
Inclusion criteria:

1. Child is aged 2 years 0 months to 7 years 11 months inclusive
2. Child has a documented diagnosis of ASD
3. Child exhibits at least one form of daily or hourly self-injurious behavior and/or aggressive behavior on the Behavior Problems Inventory - Short Form (BPI-S)71,72
4. Family lives in one of the following counties in New Mexico and Texas: Bernalillo, Santa Fe, Valencia, Sandoval, Torrance, Socorro, Cibola, Los Alamos, El Paso, Hudspeth, Otero, McKinley, San Miguel, Eddy, Chaves, or Dona Ana.
5. Caregiver is comfortable speaking and reading in English
6. The child's caregiver is at least 21 years old
7. The same caregiver is consistently available for one hour per week for a 12-week period in their home with their child between 9am and 7pm Monday through Friday to take part in the research
8. Caregiver is willing to adhere to the study intervention regimen and be willing to have a clinician come into their home for 1 hour per week for 12 weeks
9. Family lives in an area with consistent cell phone coverage

Exclusion criteria:

1. Caregiver is currently receiving ABA services or direct parent coaching to manage their child's challenging behaviors
2. Child engages in behavior that may inflict moderate to severe damage on the individual or on other people (e.g. biting through the skin, eye gouging, fracturing bones, significant damage to property) with minor or major medical intervention required.
3. Child has a sensory or physical impairment that precludes participation (e.g., epilepsy, vision or hearing impairment) or has a diagnosis of another genetic condition (e.g., fragile X syndrome)
4. Activity restrictions that limit caregiver's ability to respond to their child's challenging behaviors
5. Child has an underlying medical condition that is better treated with medical intervention
6. Child only exhibits pica at a daily or hourly frequency on the BPI-S
7. The caregiver has another child already participating in the study

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of challenging behavior | 4 week intervals
  In-session observations of challenging behavior
Parenting Stress Index | Previous 4 weeks
  Severity of parent stress

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Behavior Change Institute, Alamogordo, New Mexico

IPD SHARING:
Plan to Share IPD: No